CLINICAL TRIAL: NCT04303975
Title: An Explorative Study on the Association of High Sensitivity C-Reactive Protein (hsCRP) and Radiotherapy-Induced Toxicity in Patients With Nasopharyngeal Carcinoma
Brief Title: The Association of hsCRP and Radiotherapy-Induced Toxicity in Patients With Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jiarong Chen, MD (Other)
Responsible Party: Sponsor-Investigator, Jiarong Chen, MD, Principal Investigator, Jiangmen Central Hospital
Organization: Jiangmen Central Hospital (Other)
Other Study IDs: JM0019002
Record Dates: First submitted 2020-03-06; First posted 2020-03-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Nasopharyngeal Carcinoma; Head and Neck Cancer; Toxicity Due to Radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with neoadjuvant chemotherapy: The patients of group1 will receive one of the following treatments:
  1. neoadjuvant chemotherapy & concurrent chemoradiotherapy
  2. neoadjuvant chemotherapy & radiotherapy
  3. neoadjuvant chemotherapy & radiotherapy & adjuvant chemotherapy
  Interventions: Other: clinical measurements
- Group 2: Patients without neoadjuvant chemotherapy: The patients of group2 will receive one of the following treatments:
  1. concurrent chemoradiotherapy
  2. concurrent chemoradiotherapy & adjuvant chemoradiotherapy
  3. radiotherapy & adjuvant chemotherapy
  Interventions: Other: clinical measurements

INTERVENTIONS:
Other: clinical measurements — Only clinical parameters were recorded, no intervention was made.

SUMMARY:
The primary purpose of this study is to explore the association of high sensitivity C-reactive protein (hsCRP) and radiotherapy(RT)-induced toxicity in patients with nasopharyngeal carcinoma. In each patient, hsCRP levels in the pre- and post-RT plasma samples will be measured according to the schedule we set.

ELIGIBILITY:
Inclusion Criteria:

* Patients were pathologically newly diagnosed with nasopharyngeal carcinoma and had no previous history of other tumors
* According to the treatment strategies of doctors, patients need to receive radiotherapy with or without chemotherapy (for example, neoadjuvant chemotherapy, concurrent chemotherapy, adjuvant chemotherapy) or targeted therapy
* Willingness to sign the informed consent and return to enrolling institution for follow-up and data collection

Exclusion Criteria:

* Patients do not conform to the inclusion criteria
* Pregnant or Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* Vital organs dysfunction(for example, kidneys, heart, liver, lungs, brain)
* Other contraindications or unsuitable conditions for radiotherapy

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with nasopharyngeal carcinoma during the conducting of this trail at Jiangmen Central Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
hsCRP levels | Through treatments completion，12 weeks
  The hscrp levels in the plasma samples from each participant were measured at the following time points:
  1. at the time of diagnosis completion/before the initiation of the first neoadjuvant chemotherapy
  2. before the initiation of each neoadjuvant chemotherapy
  3. before the initiation of the first radiotherapy
  4. during radiotherapy, once a week
  5. 1 week and 4weeks after the last radiotherapy
Incidence of adverse events | Through treatments completion，12 weeks
  All adverse events were recorded during treatment(for example, oral mucositis, dermatitis).

CONTACTS AND LOCATIONS:
Overall Officials: Jiarong Chen, PhD, Principal Investigator — Affiliated Jiangmen Hospital of Sun Yat-Sen University